CLINICAL TRIAL: NCT05623657
Title: Game-Based Exercise Program and Trunk Stabilization Exercise Training in Adolescent Playing Archery
Brief Title: Comparison of the Efficiency of Game-Based Exercise Program and Trunk Stabilization Exercise Training in Adolescent Playing Archery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc. Prof., Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2022-11-12; First posted 2022-11-21 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Athlete; Itch
Keywords: Archery; trunk; balance; exergame; core stability
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk Stabilization Exercise Training Group (Experimental)
  Interventions: Other: Trunk Stabilization Exercise Training Group
- Game Based Exercise Program Group (Experimental)
  Interventions: Other: Game Based Exercise Program Group

INTERVENTIONS:
Other: Trunk Stabilization Exercise Training Group — The adolescents in this group who are involved in archery sports will be given 40 minutes of exercise training 2 days a week for 8 weeks. Exercise training will be applied as 5-10 minutes warm-up, 15-30 minutes trunk stabilization exercises, 5-10 minutes cooling down, and stretching exercises. The number of repetitions and difficulty levels of the exercises will gradually increase in the 3rd and 6th weeks.
  Arms: Trunk Stabilization Exercise Training Group
Other: Game Based Exercise Program Group — At least 4 different games selected from Xbox 360 Kinect® games will be applied to adolescents practicing archery sports in this group for a total of 40 minutes with the physiotherapist. The games will be selected from games that include movement patterns similar to the exercises of the trunk stabilization exercise group. Game-based exercise training is planned to be performed twice a week for a total of 8 weeks.
  Arms: Game Based Exercise Program Group

SUMMARY:
The aim of our study is to investigate the effects of a game-based exercise (Exergame) program and trunk stabilization exercise training on shooting performance, reaction time, trunk muscle endurance and balance in adolescents playing archery. While the importance of the effect of trunk stabilization on shooting performance is mentioned in individuals practicing archery, it is emphasized that trunk stabilization training increases sportive performance and protects against injuries in individuals interested in sports for the upper extremity. However, no study is found that directly compared game-based exercise programs and trunk stabilization exercise training in adolescents who play archery. Therefore, two different training programs will be given to the adolescents playing archery at the Archers Foundation Sports Club in Istanbul, and Shooting performance, reaction time, trunk muscle endurance, and balance levels will be evaluated before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Archers who have been practicing archery for at least 1 year
* Roller or Olympic archers

Exclusion Criteria:

* Archers with a history of musculoskeletal injuries causing physical limitation in the last 6 months.
* Archers who did not volunteer to participate in the study.
* Archers with any visual and hearing disabilities.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Core Endurance Tests | Change from baseline to 8 weeks
  McGill's tests will be used to examine participants' core endurance. These tests consist of four positions: the trunk anterior flexor test, the right and left lateral plank, and the trunk posterior extensor test. Participants will perform one practice trial that will last a few seconds to confirm position and then one actual test trial will be recorded per position where the maximum time (seconds) participants could hold a static position was measured. The same investigator visually will determine the end of all tests.
Star Excursion Balance Test (SEBT) : | Change from baseline to 8 weeks
  The test requires strength, flexibility, and proprioception. It is a measure of dynamic balance that provides a significant challenge to athletes and physically active individuals. The participant performing the test must maintain their balance on one leg while using the other leg to reach as far as possible in 8 different directions. The participant (standing on his/her left leg for example) must reach in 8 different positions, once in each of the following directions: anterior, anteromedial, medial, posteromedial, posterior, posterolateral, lateral and anterolateral. The anterior, posteromedial and posterolateral directions appear to be important to identify individuals with chronic ankle instability and athletes at greater risk of lower extremity injury.
Reaction Time Evaluation: | Change from baseline to 8 weeks
  It plans to use the free platform game (Reaction Time) available in the Android app. Test The test is performed using a tablet in a quiet and lighted room, the tablet will be placed on the desktop with a stabilizing stand.Athletes participating in the study will be asked to sit in a chair so that they are comfortable on the table.Test protocols after a verbal explanation, the athletes will be given one trial before the reaction time measurement. Stimuli given 5 times at fixed and random intervals, the average of the 5 trials results in the reaction time in milliseconds.
  The participant is asked to touch the middle of the tablet screen with his finger when the blue color appears.When the green color appears, the screen continues to be touched, and when the green color appears, the screen is quickly stopped being touched. All athletes have a dominant and The non-dominant side uses the hands, index fingers.

SECONDARY OUTCOMES:
Shooting Performance Evaluation: | Change from baseline to 8 weeks
  Outdoor Shooting Performance: A total of 72 arrows, 2 x 36 arrows, will be shot at the distances specified by the International Archery Federation. The series were shot as 6 arrows each. A total of 360 points will be calculated. The higher the score, the better the performance of the athlete. Each athlete used his/her own bow and arrow, and the athlete must complete the shots within certain time limits.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No